CLINICAL TRIAL: NCT07346248
Title: Postoperative Complications After Neoadjuvant Chemoradiotherapy or Short-course Radiotherapy and Total Neoadjuvant Treatment: a Multicentric Retrospective Cohort Study
Acronym: POCAT
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 5019
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Adult Patients With Locally Advanced Rectal Cancer Indicated to Neoadjuvant Therapy and Surgery
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemoradiotherapy: Patient received chemoradiotherapy or short course radiotherapy before surgery
  Interventions: Procedure: Chemoradiotherapy
- TNT: TNT neoadjuvant treatment
  Interventions: Procedure: Chemoradiotherapy

INTERVENTIONS:
Procedure: Chemoradiotherapy — Comparing

SUMMARY:
The primary objective of the study is to compare the rate of postoperative complications between rectal cancer patients undergoing standard neoadjuvant chemoradiotherapy or short- course radiotherapy and patients receiving TNT. The secondary objectives of the study include the evaluation of treatment-related adverse reactions and postoperative complications in elderly patients receiving the treatments and the comparison of treatment-related adverse reactions and postoperative complications in patients receiving induction versus consolidation TNT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced (T2N+, T3N+, T4N0, or T4N+) rectal adenocarcinoma who underwent neoadjuvant chemoradiotherapy or short-course radiotherapy or TNT and surgery between January 2016 and January 2025;
* Patients who underwent restorative or non-restorative surgery;
* Patients undergoing open, laparoscopic, or robotic intervention.

Exclusion Criteria:

* Patients who underwent non-operative management after neoadjuvant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all consecutive adult patients with locally advanced rectal adenocarcinoma who started a classical neoadjuvant or short-course radiotherapy or TNT treatment between January 2016 and January 2025 at the investigational centers.
Sampling Method: Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
90 days postoperative complications | 12 months
  The primary endpoint of the study is the rate of 90-day postoperative complications between the study cohorts.
The primary endpoint of the study is the rate of 90-day postoperative complications between the study cohorts. | 3 months
  The primary endpoint of the study is the rate of 90-day postoperative complications between the study cohorts.

SECONDARY OUTCOMES:
90 days severe postoperative complications between the cohorts | 12 months
  The rate of 90-day severe postoperative complications between the study cohorts.
90-day Comprehensive Complication Index | 12 months
  The median of the 90-day Comprehensive Complication Index (CCI) between the study cohorts.
Treatment-related adverse reactions | 12 months
  The rate of treatment-related adverse reactions between the study cohorts.
Severe treatment-related adverse reactions | 12 months
  The rate of severe treatment-related adverse reactions between the study cohorts.
90-day postoperative complications between patients receiving neoadjuvant chemoradiotherapy,short-course radiotherapy, induction TNT, and consolidation TNT. | 12 months
  The rate of 90-day postoperative complications between patients receiving neoadjuvant chemoradiotherapy,short-course radiotherapy, induction TNT, and consolidation TNT.
Treatment-related adverse reactions between patients receiving neoadjuvant chemoradiotherapy,short-course radiotherapy, induction TNT, and consolidation TNT | 12 months
  The rate of treatment-related adverse reactions between patients receiving neoadjuvant chemoradiotherapy,short-course radiotherapy, induction TNT, and consolidation TNT.
The rate of 90-day postoperative complications between the two cohorts in a sub-population of elderly patients | 12 months
  The rate of 90-day postoperative complications between the two cohorts in a sub-population of elderly patients (≥ 70 years old at the time of diagnosis).
The rate of treatment-related adverse reactions between the study cohorts in a sub-population of elderly patients | 12 months
  The rate of treatment-related adverse reactions between the study cohorts in a sub-population of elderly patients (≥ 70 years old at the time of diagnosis).

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, Surgery, PhD, Study Director — Director Colon and Rectal Surgery -Director General Surgery Residency Program - Co-Director IBD Center Humanitas Research Hospital / Humanitas University
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No